CLINICAL TRIAL: NCT05339854
Title: Evaluation of Cardio-pulmonary, Physcial and Neuro-psychiatric Function in Patients Who Survived a Therapy-refractory Cardiac Arrest With Extracorporeal Cardiopulmonary Resuscitation.
Brief Title: Evaluation of eCPR Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Düsseldorf (Other)
Responsible Party: Principal Investigator, Tharusan Thevathasan, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ECPR Outpatient Clinic
Record Dates: First submitted 2022-04-10; First posted 2022-04-21 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation; Extracorporeal Membrane Oxygenation Complication; Myocardial Infarction; Cardiogenic Shock
MeSH Terms: conditions — Heart Arrest; Myocardial Infarction; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood draw: Sodium, Potassium, Chloride, Calcium, Magnesium, Creatinine, Urea, Uric acid, Bilirubin, Cholesterol (total, HDL, LDL), Triglyceride, Lipoprotein (a), HbA1c, NT-proBNP, Creatinkinase (CK), CK-MB, Myoglobin, ALT, AST, Gamma-GT, Alkaline phosphatase, GLDH, Lipase, LDH, CRP, Procalcitonin, Albumin, Iron, Ferritin, Transferrin, Transferrin saturation, Haptoglobin, Free hemoglobin, Complete blood count, Quick, PTT, TSH, T4, T3, Cortisol, venous arterial blood gas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECPR survivor: Adult patient who survived therapy-refractory cardiac arrest with extracorporeal cardiopulmonary resuscitation (ECPR).

SUMMARY:
A cardiac arrest event has severe impact on the patient´s health-related quality of life. Survival of cardiac arrest does not innately translate to favorable quality of life. In particular, highly invasive resuscitation strategies, including extracorporeal cardio-pulmonary resuscitation (ECPR) due to therapy-refractory cardiac arrest, may have impact on long-term outcomes. Therefore, apart from acute medical treatment and physical rehabilitation, long-term effects on cardio-pulmonary, physical and neuro-psychiatric functions after cardiac arrest survival have to be evaluated and optimized. We plan to investigate a bundle of cardio-pulmonary, physical and neuro-psychiatric functions in patients who survived a therapy-refratory cardiac arrest with ECPR.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Survival of cardiac arrest
* Use of extracorporeal cardiopulmonary resuscitation (ECPR) with veno-arterial extracorporeal membrane oxygenation (VA-ECMO) or ECMELLA (VA-ECMO and left-ventricular Impella micro-axial pump)

Exclusion Criteria:

* Non-adult patients
* No cardiac arrest
* No use of ECPR
* Inability to comply with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who suffered from cardiac arrest and were treated with ECPR.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | LVEF witihin one year after index cardiac arrest event.
  LVEF measured with transthoracic echocardiography.

SECONDARY OUTCOMES:
Cognitive function | Cognitive function witihin one year after index cardiac arrest event.
  Cognitive function measured with a standardized questionnaire and following established scores:
  1. Mini-mental-status-test [0-30 points; higher score means better outcome],
  2. Cerebral Performance Categories Scale [1-5; lower score means better outcome].
Sign and symptoms of heart failure | Sign and symptoms of heart failure witihin one year after index cardiac arrest event.
  Sign and symptoms of heart failure measured with a standardized questionnaire and following established score: European Quality of Life 5 Dimensions 3 Level Version [0-100 points; higher score means better outcome].
Activity of daily living (ADL) | ADL witihin one year after index cardiac arrest event.
  ADL measured with a standardized questionnaire and following estbalished score:
  Barthel index [0-100 points; higher score means better outcome].
Comorbidity level | Comorbidity level witihin one year after index cardiac arrest event.
  Comorbidity level measured with following established score: Charlson comorbidity index [0-24 points; lower score means better outcome].
Number of cardiovascular medications | Number of cardiovascular medication witihin one year after index cardiac arrest event.
  Number of cardiovascular medications documented with a standardized questionnaire.
Cardiac stress test: Ergometry | Physical function witihin one year after index cardiac arrest event.
  Quantitative test to evaluate cardiopulmonary exercise tolerance and physical capacity by using a bicycle.
Cardiac stress test: Walking distance | Physical function witihin one year after index cardiac arrest event.
  Quantitative test to evaluate endurance and aerobic capacity by walking for six minutes (six minute walk test).
Vital function: Blood pressure | Blood pressure witihin one year after index cardiac arrest event.
  Non-invasive blood pressure measurement at rest (unit: mmHg).
Vital function: Electrocardiogram (ECG) | ECG activity witihin one year after index cardiac arrest event.
  12-lead ECG measurement at rest.
Vital function: Peripheral oxygen saturation | Peripheral oxygen saturation witihin one year after index cardiac arrest event.
  Peripheral oxygen saturation measurement at rest by using pulsoximetry (unit: percent).

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skurk, MD, Study Director — Charite Univesity; Tharusan Thevathasan, MD, Principal Investigator — Charite Univesity
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No